CLINICAL TRIAL: NCT06010680
Title: Phase I Clinical Trial of Substance Balance of [14C]SHR2554 in Healthy Chinese Subjects
Brief Title: A Study to Evaluate the Mass Balance of [14C]SHR2554 in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SHR2554-I-111
Record Dates: First submitted 2023-08-20; First posted 2023-08-24 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Intervention Model Description: Single oral dose of [14C]SHR2554
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [14C]SHR2554 (Experimental)
  Interventions: Drug: [14C]SHR2554

INTERVENTIONS:
Drug: [14C]SHR2554 — Patients will receive single dose of orally [14C]SHR2554 on Day 1.

SUMMARY:
Evaluate the Mass Balance of [14C]SHR2554 in Healthy Adult Male Volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult males between 18 and 45 years;
2. Total Body weight ≥50 kg, and the body mass index (BMI) of 19 to 26 kg/m2;
3. Sign the informed consent form prior to the trial and have a full understanding of the trial's procedures, content, and potential adverse reactions;
4. Ability to communicate effectively with the researchers and comply with the trial requirements.

Exclusion Criteria:

1. Comprehensive physical examination, vital signs, laboratory tests, 12-lead ECG, chest X-ray (posteroanterior), anal digital examination, abdominal ultrasound with clinically significant abnormalities as determined by the investigator;
2. Resting corrected QT interval (QTcF) >450 ms as obtained from the 12-lead ECG (Note: QTcF interval must be calculated according to Fridericia's method);
3. Positive results in any of the following tests: hepatitis B surface antigen or hepatitis B e antigen, hepatitis C virus antibodies or HIV antigen/antibody combination test (HIV-Ag/Ab);
4. Clinically significant abnormalities in ophthalmic examination (slit lamp, intraocular pressure, and fundus photography);
5. Have taken any clinical trial drug or participated in any clinical trial within 3 months before administration;
6. CYP3A4 inducers or inhibitors were taken within 30 days before administration;
7. Have taken any prescription or over-the-counter drugs, vitamin products, health care drugs or traditional Chinese medicines within 14 days before administration;
8. History of any clinically significant medical conditions or conditions that the investigator deems may affect the trial results, including but not limited to cardiovascular, respiratory, endocrine, nervous, digestive, urinary, immune, mental, and metabolic diseases;
9. History of organic heart disease, congestive heart failure, myocardial infarction, angina pectoris, unexplained history of arrhythmia, history of torsades de pointes, history of ventricular tachycardia, atrioventricular conduction block, history of QT prolongation syndrome, or family history of QT prolongation syndrome (confirmed by genetic testing or sudden cardiac death in a close relative at a young age due to cardiac reasons);
10. Those who have undergone major surgery within 6 months before administration or that surgical incision has not completely healed; Major surgery includes, but is not limited to, any surgery that is at significant risk of bleeding, prolongs the period of general anesthesia, or has an incision biopsy or significant traumatic injury;
11. Hemorrhoids or anal diseases accompanied by regular/ongoing rectal bleeding; inability to swallow or a history of gastrointestinal dysfunction such as irritable bowel syndrome, inflammatory bowel disease, or previous gastric resection surgery that may affect drug absorption as determined by the investigator;
12. Allergic predisposition, such as known history of allergy to two or more substances; or deemed by the investigator to be potentially allergic to the investigational drug or its excipients;
13. Habitual constipation or diarrhea;
14. History of alcoholism with alcohol consumption over 14 units per week; and can't abstain from smoking and alcohol during the study;
15. Heavy smoker or habitually use nicotine-containing products;
16. Have a history of drug abuse or have used soft drugs (such as: marijuana) within 3 months before administration or take drugs (such as cocaine, amphetamines, phencyclidine, etc.) within 1 year before administration; or positive urine drug abuse test during screening periods;
17. Habitual consumption of grapefruit juice or excessive tea, coffee and/or caffeinated beverages (more than 8 cups a day, 1 cup = 250 mL) and unable to quit during the study period;
18. Those who cannot tolerate venipuncture or with a history of needle-sickness and blood-sickness;
19. Workers who require long-term exposure to radioactive conditions; or those who have significant radiation exposure (≥ 2 chest/abdominal CT scans, or ≥3 other X-ray tests) within 1 year prior to administration or who have participated in radiopharmaceutical labeling tests;
20. Blood donation no less than 400 mL or have blood transfusion within 3 months of dosing;
21. Vaccination within one month prior to screening or planning to be vaccinated during the trial;
22. Intention to conceive or donate sperm during the trial period or within one year after completing the trial, or refusal to strictly adhere to contraceptive measures by the participant and their spouse/partner from the time of signing the informed consent form until one year after completing the trial;
23. Subjects who, in the opinion of the Investigator should not participate in this study.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2023-10-07 (Actual); Primary Completion 2023-11-27 (Actual); Study Completion 2023-11-27 (Actual)

PRIMARY OUTCOMES:
Cumulative recovery and recovery rate of total radioactive substance in urine and feces | 0-288 hours
Percentage of parent drug and its metabolites in plasma as a percentage of total radioactive exposure (%AUC) | 0-240 hours
Percentage of parent drug and its metabolites in urine and feces as a percentage of administered dose (%Dose) | 0-288 hours
Radioactivity Tmax | 0-240 hours
Radioactivity Cmax | 0-240 hours
Radioactivity AUC | 0-240 hours
Radioactivity t1/2 | 0-240 hours
Radioactivity CL/F | 0-240 hours
Radioactivity Vz/F | 0-240 hours
1Total radioactivity ratio for blood/plasma | 0-72 hours

SECONDARY OUTCOMES:
Plasma SHR2554: Tmax | 0-240 hours
Plasma SHR2554: Cmax | 0-240 hours
Plasma SHR2554: AUC | 0-240 hours
Plasma SHR2554: t1/2 | 0-240 hours
Plasma SHR2554: CL/F | 0-240 hours
Plasma SHR2554: Vz/F | 0-240 hours
Plasma SHR2554: λz | 0-240 hours
AEs and SAEs | 0-12 days

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Suzhou University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided